CLINICAL TRIAL: NCT06499545
Title: Plantar Pressures After Pressure Release of the Flexor Digitorum Brevis Muscle Versus a Non-emission Laser: Clinical Trial.
Brief Title: Plantar Pressures After Pressure Release of the Flexor Digitorum Brevis Muscle Versus a Non-emission Laser.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Physiotherapist responsible area, Mayuben Private Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1912202200923 B
Record Dates: First submitted 2024-07-07; First posted 2024-07-12 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Manual Therapy; Myofascial Pain Syndrome; Foot; Flat Foot
MeSH Terms: conditions — Myofascial Pain Syndromes; Flatfoot | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pressure release (Experimental): Application of pressure release as a trigger point treatment of the flexor digitorum brevis muscle. Performing 3 pressure cycles until the disappearance of the referred pain for a minimum of 90 seconds.
  Interventions: Other: Pressure release
- Non-emision Laser (Sham Comparator): Application of a non-emitting laser for 5 minutes.
  Interventions: Other: Non emision Laser

INTERVENTIONS:
Other: Pressure release — Release of pre-pressure at the latent trigger point of flexor digitorum brevis
  Arms: Pressure release
Other: Non emision Laser — Non emision laser in Flexor digitorum brevis latent trigger point
  Arms: Non-emision Laser

SUMMARY:
In this study we will test the effects of pressure release on the Flexor digitorum brevis muscle on the plantar pressures variables using a pressure platform.

ELIGIBILITY:
Inclusion criteria:

* Participants who came to the clinic presenting with pain in both heels and who were diagnosed with active or latent myofascial trigger point in bilateral flexor digitorum brevis muscles.
* Myofascila trigger points of flexor digitorum brevis were the only ones diagnosed in the foot.
* All participants with normal body mass, without obesity.

Exclusion criteria:

* Diagnosis of lower limb injury, such as plantar fasciitis, tendinopathy, bursitis, ligamentous injuries.
* History of previous lower limb surgery.
* Participants will not be subjected to ankle stretching or any other treatment.
* Diabetes due to possible elevation of plantar pressure.
* Toe deformities such as hammertoes and hallux valgus due to possible alteration of plantar pressure.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-08-03 (Actual)

PRIMARY OUTCOMES:
Variables of plantar pressures with platform before non-emission laser | Through study completion, an average of 2 days
  For 30 seconds we will record the plantar pressure variables in grams per square centimetre.
Variables of plantar pressures with platform before pressure release | Through study completion, an average of 2 days
  For 30 seconds we will record the plantar pressure variables in grams per square centimetre.
Variable footprint planting surface with platform before non-emission laser | Through study completion, an average of 2 days
  For 30 seconds we will record the area of the footprint in square centimetres.
Variable footprint plantar surface with platform before pressure release | Through study completion, an average of 2 days
  For 30 seconds we will record the plantar pressure variables in grams per square centimetre.
Variables of plantar pressures with platform after non-emission laser | Through study completion, an average of 2 days
  For 30 seconds we will record the plantar pressure variables in grams per square centimetre.
Variables of plantar pressures with platform after preassure release | Through study completion, an average of 2 days
  For 30 seconds we will record the plantar pressure variables in grams per square centimetre.
Variable footprint planting surface with platform after non-emission laser | Through study completion, an average of 2 days
  For 30 seconds we will record the area of the footprint in square centimetres.
Variable footprint planting surface with platform after pressure release | Through study completion, an average of 2 days
  For 30 seconds we will record the area of the footprint in square centimetres.

CONTACTS AND LOCATIONS:
Overall Officials: Eva María Martínez-Jiménez, PhD, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Mayuben Clinic, San Sebastián de los Reyes, Madrid, Spain